CLINICAL TRIAL: NCT03138525
Title: Immune Profiling During Ocrelizumab Treatment in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Howard L Weiner, Director, Partners Multiple Sclerosis Center; Co-Director, Ann Romney Center for Neurologic Diseases, Brigham and Women's Hospital
Other Study IDs: ML39789
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis; Healthy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Subjects with multiple sclerosis (MS) initiating treatment with ocrelizumab
  Interventions: Other: Blood sampling (MS)
- Healthy: Healthy individuals serving as controls to the subjects with MS
  Interventions: Other: Blood sampling (controls)

INTERVENTIONS:
Other: Blood sampling (MS) — Blood samples will be collected before initiation of Ocrelizumab treatment and after 6 and 12 months of treatment.
  Groups: Multiple Sclerosis
Other: Blood sampling (controls) — Blood samples will be collected once at enrollment.
  Groups: Healthy

SUMMARY:
The purpose of this study is to assess effects of B cell depletion on the immune system in patients with relapsing forms of multiple sclerosis (MS) treated with ocrelizumab. This will be done by collecting blood from patients starting treatment with ocrelizumab before the first infusion and before the infusions at 6 and 12 months. The effects on the immune system will be assessed by performing transcriptome profiling of immune cells, measuring serum levels of microRNAs, and analyzing serum autoantibody immune signatures using antigen arrays. In addition, blood will be collected once from a group of healthy individuals to serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing form of MS starting treatment with ocrelizumab at Partners MS Center
* Healthy controls
* Ability to understand and sign informed consent

Exclusion Criteria - All subjects:

* Other concomitant autoimmune or inflammatory diseases
* Ongoing treatment with other immunomodulatory medications
* Previous treatment with rituximab, methotrexate, cyclophosphamide, mitoxantrone, mycophenolate mofetil, or alemtuzumab
* Pregnancy or lactation
* Hypersensitivity to ocrelizumab

Exclusion Criteria - Healthy Controls:

* MS
* First-degree relatives with MS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with relapsing form of MS starting treatment with ocrelizumab at Partners MS Center
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Monocyte Transcriptome Profiling | 12 months
  Changes in messenger ribonucleic acid (mRNA) expression
Antigen microarrays | 12 months
  Changes in serum autoantibody immune signatures
Serum microRNA profiles | 12 months
  Changes in serum microRNA expression

CONTACTS AND LOCATIONS:
Overall Officials: Howard L Weiner, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States